CLINICAL TRIAL: NCT05694676
Title: Relationship Between Prenatal Maternal Depression and Anxiety and the Quality of General Movements of Healthy Term Infants at 3 Months
Brief Title: Relationship Between Prenatal Maternal Distress and the Quality of General Movements at 3 Months
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aynur Başaran, MD, Prof, Karamanoğlu Mehmetbey University
Other Study IDs: 11-2022/02
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy; Infant Development; Maternal Distress
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers: Mothers aged 18 to 40 years, who have singleton pregnancy.
  Interventions: Other: State-Trait Anxiety Inventory-Trait, (STAI-T); Other: Beck Depression Inventory, (BDI)
- Infants: Infants were born at 36-42 weeks of gestation without complication.
  Interventions: Other: Assessment of the quality of Genaral Movements (GMs)

INTERVENTIONS:
Other: Assessment of the quality of Genaral Movements (GMs) — The variation, complexity and fluency of movements over a video recording is done and the quality of GMs is classified as normal-optimal, normal-suboptimal, mildly abnormal, and definitely abnormal movements.
  Other Names: Prechtl's General movements (GMs)
  Groups: Infants
Other: State-Trait Anxiety Inventory-Trait, (STAI-T) — The scale consists of 20 items in total and provides a four-point Likert type measurement (1- anxiety symptom is not present, 4- the symptom lasts all the time). Scores range from 20 (low anxiety) to 80 (high anxiety).
  Groups: Mothers
Other: Beck Depression Inventory, (BDI) — BDI contains 21 items and rates the depressive symptoms for the last week. Each item has four options and is scored between 0 and 3. The total score ranges from 0 to 63. Higher scores indicate more severe depression
  Groups: Mothers

SUMMARY:
Depression and anxiety symptoms are common during pregnancy which may disturb the intrauterine environment by affecting the mother's physiological responses to stress, and ultimately impair fetal and postnatal development. There is increasing evidence about the effects of maternal distress on young brain tissue leading to some structural changes. The neurological footprints of these structural changes on the young brain may be caught early in life by a video assessment of General Movements (GMs) quality.

DETAILED DESCRIPTION:
Depression and anxiety symptoms are common during pregnancy and are estimated to affect 7% - 20% of pregnant women, constituting significant risks for mothers and babies. Depression and anxiety may disturb the intrauterine environment by affecting the mother's physiological responses to stress, and ultimately impair fetal and postnatal development. Increasing evidence shows that prenatal exposure to maternal depression and anxiety is associated with several lifelong adverse outcomes in children, including physical health problems, emotional and behavioral difficulties, and low verbal IQ.

Such maladaptive outcomes are thought to have a neurobiological basis and there is increasing evidence about the effects of maternal distress on young brain tissue leading to some structural changes. However, what is more important is that the neurological footprints of these structural changes on the young brain can be caught early in life. The neurological status of infants can be determined early in life by video assessment of General Movements (GMs) quality. In this study at the age of 3 months, a video assessment of the quality of GMs will be performed to evaluate neurologic conditions.

ELIGIBILITY:
Mothers Inclusion Criteria:

* Mothers aged 18 to 40 years,
* Singleton pregnancy
* No smoking during prengnancy
* No illicit drug or alcohol use during pregnancy,
* No major health conditions requiring invasive treatments (e.g., dialysis, blood transfusions, chemotherapy),
* No diagnosis of psychotic illnesses (eg, schizophrenia,bipolar or borderline personality disorder), and
* No major autoimmune diseases
* No pregnancy-related complications: (including prenatal infection, pregnancy-included hypertension, gestational diabetes, oligohydramnios, polyhydramnios, preterm labor, vaginal bleeding, placenta previa, or anemia).

Infant inclusionary criteria:

* infants were born at 36-42 wk of gestation
* uncomplicated singleton birth,
* no pre-existing neurologic conditions or major head trauma, neonatal intensive care unit stay limited to observation only (ie, no interventions), and
* infant discharged from the hospital with the mother.

Mothers Exclusion Criteria:

* post partum depression and/or anxiety
* delivery complication

Infant exclusion criteri:

* infant birth before 36 weeks gestation
* infant weight lower 2500gr at birth
* Apgar score 0f <7 at 5 minutes
* Major neonatal complications
* Identified neurologic, genetic or congenital syndrome

Ages: 10 Weeks to 20 Weeks | Sex: All
Age Groups: Child
Study Population: Mothers aged 18 to 40 years, who have singleton pregnancy.
  Infants were born at 36-42 weeks of gestation without complication.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Relationship Between Prenatal Maternal Anxiety and the Quality of General Movements | 3-5 months
  Univariate statistical analyses will be performed to calculate differences in mothers' STAI-T scores between children with normal and abnormal GMs.
Relationship Between Prenatal Maternal Depression and the Quality of General Movements | 3-5 months
  Univariate statistical analyses will be performed to calculate differences in mothers' BDI scores between children with normal and abnormal GMs.

SECONDARY OUTCOMES:
Multivariate analyses will be carried out with control variables | 3-5 months
  Significant primary outcome measures will be controlled with:
  * Maternal age (years)
  * Maternal education (Literate, Elementary school, Middle School, High school, University)
  * Marital status (married, separated, divorced, widow)
  * Maternal height (m)
  * Maternal weight before pregnancy (kg)
  * Maternal weight at birth (kg)
  * Maternal BMI before pregnancy (Maternal weight before pregnancy/Maternal height) (kg/m^2)
  * Maternal BMI at birth (Maternal weight at birth/Maternal height)(kg/m^2)
  * Type of delivery (Vaginal spontaneous, Instrumental, Assisted vaginal, Elective C/S, Emergency C/S),
  * Birth order
  * Gestational age at birth (days)
  * Infant birth weight (grams)
  * Infant birth height (cm)
  * Infant birth head circumference (cm)
  * Infant gender (boy, girl)
  * Infant 1st and 5th minute Apgar scores
  * Breastfeeding (>6wk, <=6 wk)

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Basaran, MD,Prof, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)